CLINICAL TRIAL: NCT01088672
Title: Thrombectomy REvascularization of Large Vessel Occlusions in Acute Ischemic Stroke (TREVO)
Acronym: TREVO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Stryker Neurovascular (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DQR0036
Record Dates: First submitted 2010-03-15; First posted 2010-03-17 (Estimated); Results first posted 2015-07-17 (Estimated); Last update posted 2015-07-17 (Estimated); Status verified 2015-07

CONDITIONS: Ischemic Stroke
Keywords: Stroke; Ischemic; Thrombus; Embolectomy; Thrombectomy; Concentric; Embolus; Mechanical; Trevo
MeSH Terms: conditions — Ischemic Stroke; Stroke; Ischemia; Thrombosis; Embolism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Acute Ischemic Stroke (Other): Single arm post market surveillance study for CE marked mechanical thrombectomy device, Trevo retriever for treatment of eligible patients experiencing acute ischemic stroke Mechanical thrombectomy intervention for all subjects in Acute Ischemic Stroke
  Interventions: Procedure: Mechanical Thrombectomy

INTERVENTIONS:
Procedure: Mechanical Thrombectomy — The Trevo device is intended to restore blood flow in the neurovasculature by removing thrombus in patients experiencing ischemic stroke.
  Other Names: Trevo Procedure

SUMMARY:
To determine the revascularization rate of the CE-marked Trevo device in large vessel occlusions in ischemic stroke patients.

* Revascularization, defined as at least TICI 2a in the vascular territory treated at end of the neuro interventional procedure.

DETAILED DESCRIPTION:
* Clinical outcomes at 90 days
* Mortality at 90 days
* Device-related serious adverse events (DRSAEs)
* Symptomatic ICH rate within 24 (-6/+12) hours post-procedure

ELIGIBILITY:
Inclusion Criteria:

* Age 18-79 (has had 18th birthday, but not yet had 80th birthday)
* NIHSS 8 - 30
* Anticipated life expectancy of at least 6 months
* No significant pre-stroke disability (mRS less than or equal to 1)
* Written informed consent to participate given by patient or legal representative
* Angiographic confirmation of a persistent large vessel occlusion, in the internal carotid, middle cerebral M1 and/or M2 segments, basilar or vertebral arteries
* Treatable within 8 hours of symptom onset, defined as the first pass being made with the Trevo device.

Exclusion Criteria:

* Baseline glucose of < 50 mg/dL (2.78 mmol) or > 400 mg / dL (22.20 mmol)
* Known hemorrhagic diathesis, coagulation factor deficiency, or oral anticoagulant therapy with INR > 3.0
* Treated with Heparin within 48 hours with a PTT greater than 2 times the lab normal
* Baseline platelet count < 30,000
* History of severe allergy (more than rash) to contrast medium
* Severe, sustained hypertension (SBP > 185 mm Hg or DBP > 110 mm Hg) NOTE: If the blood pressure can be successfully reduced and maintained at the acceptable level using medication (i.e. Nipride), the patient can be enrolled
* Woman of child bearing potential who is known to be pregnant
* Patient participating in another clinical study or protocol
* For anterior circulation strokes: strokes involving greater than 1/3 of the MCA territory, as determined by hypodensity on the baseline non- contrast CT, or low CBV on CT Perfusion imaging, or restricted diffusion on DWI images
* For posterior circulation strokes within the midbrain and/or pons, extensive hypodensity on the baseline CT, or low CBV on CT Perfusion imaging, or extensive restricted diffusion on DWI images
* Baseline CT/MR evidence of significant mass effect with midline shift
* Baseline CT/MR evidence of hemorrhage
* Baseline CT/MR evidence of intracranial tumor (except small meningioma)
* Angiographic evidence of vasculitis or arterial dissection
* High grade stenosis that cannot be treated safely or which prevents access to the thrombus with the Trevo device
* Angiographic evidence of excessive arterial tortuosity that precludes the Trevo device from reaching the thrombus

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-02; Primary Completion 2011-08 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nils Wahlgren, MD, Principal Investigator — Karolinska University Hospital in Solna; Olav Jansen, MD, Principal Investigator — Universitätsklinikum Schleswig-Holstein - Campus Kiel UK S-H
Locations (7):
- Christian Doppler Clinic, Salzburg, Austria
- Germany (3):
  - Universitätsklinik Göttingen, Göttingen
  - University Hospital Schleswig-Holstein Campus Kiel, Kiel
  - Technische Universität München, Munich
- Spain (2):
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital Universitari Germans Trias i Pujols, Barcelona
- Karolinska University Hospital, Stockholm, Sweden

REFERENCES:
- [Result] Jansen O, Macho JM, Killer-Oberpfalzer M, Liebeskind D, Wahlgren N; TREVO Study Group. Neurothrombectomy for the treatment of acute ischemic stroke: results from the TREVO study. Cerebrovasc Dis. 2013;36(3):218-25. doi: 10.1159/000353990. Epub 2013 Oct 12. PMID 24135533
- [Derived] Shi ZS, Liebeskind DS, Xiang B, Ge SG, Feng L, Albers GW, Budzik R, Devlin T, Gupta R, Jansen O, Jovin TG, Killer-Oberpfalzer M, Lutsep HL, Macho J, Nogueira RG, Rymer M, Smith WS, Wahlgren N, Duckwiler GR; Multi MERCI, TREVO, and TREVO 2 Investigators. Predictors of functional dependence despite successful revascularization in large-vessel occlusion strokes. Stroke. 2014 Jul;45(7):1977-84. doi: 10.1161/STROKEAHA.114.005603. Epub 2014 May 29. PMID 24876082

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Acute Ischemic Stroke
Started | 60
Completed | 60
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Acute Ischemic Stroke
Number analyzed (Participants) | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.7 (13.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33
  Male | 27
Region of Enrollment [Number; unit: participants]
  Spain | 22
  Austria | 16
  Germany | 19
  Sweden | 3
NIHSS [Mean (Standard Deviation); unit: units on a scale] — The National Institutes of Health Stroke Scale, or NIH Stroke Scale (NIHSS) is a tool used by healthcare providers to objectively quantify the impairment caused by a stroke. The maximum (worst) possible score is 42, with the minimum (best) score being a 0.
  http://en.wikipedia.org/wiki/Nihss
  units on a scale | 17.7 (4.8)

OUTCOME MEASURES:

1. Primary Outcome: Revascularization Status
Description: Revascularization, defined as at least TICI 2a in the vascular territory treated at end of the neuro interventional procedure
  Thrombolysis in Cerebral Infarction (TICI) grading system for perfusion (ie blood flow through a vessel) Grade 0:No Perfusion. No antegrade flow beyond the point of occlusion. Grade 1:Penetration With Minimal Perfusion. Grade 2:Partial Perfusion. Grade 2a:Only partial filling (<2/3) of the entire vascular territory is visualized.
  Grade 2b:Complete filling of all of the expected vascular territory is visualized, but slower ...
  Grade 3:Complete Perfusion. For complete info see Higashida RT, Furlan AJ, Roberts H, Tomsick T, Connors B et al. (2003) Trial design and reporting standards for intra-arterial cerebral thrombolysis for acute ischemic stroke. Stroke 34: e109-e137.10.1161/01.STR.0000082721.62796.09 PubMed: 12869717[PubMed]
Time Frame: Post-procedure, immediate=at the end of the procedure, per last angiogram during treatment
Measure: Number; unit: percentage of subjects TICI 2 or >
Arm/Group | Acute Ischemic Stroke
Number analyzed (Participants) | 60
percentage of subjects TICI 2 or > | 92

2. Secondary Outcome: Clinical Outcomes at 90 Days
Description: Good clinical outcome is defined as an modified Rankin Scale (mRS) score of 0-2 at 90 days.
  mRS 0-2 indicates functional independence 0 - No symptoms.
  1. - No significant disability. Able to carry out all usual activities, despite some symptoms.
  2. - Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities.
  3. - Moderate disability. Requires some help, but able to walk unassisted.
  4. - Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted.
  5. - Severe disability. Requires constant nursing care and attention, bedridden, incontinent.
  6. - Dead.
  https://en.wikipedia.org/wiki/Modified_Rankin_Scale
Time Frame: 90-day
Measure: Number; unit: percentage of subjects with mrs 0-2
Arm/Group | Acute Ischemic Stroke
Number analyzed (Participants) | 60
percentage of subjects with mrs 0-2 | 55

3. Secondary Outcome: Mortality at 90 Days
Description: All cause mortality through 90 days post procedure.
Time Frame: 90-day
Measure: Number; unit: participants
Arm/Group | Acute Ischemic Stroke
Number analyzed (Participants) | 60
participants | 12

ADVERSE EVENTS:
Time Frame: 90 days
Description: All events adjudicated by CEC
Arm/Group | Acute Ischemic Stroke
Serious Adverse Events (participants affected / at risk) | 12/60
Other Adverse Events (participants affected / at risk) | 3/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Acute Ischemic Stroke (N=60)
Death (Vascular disorders) | 12 (12)
SICH (Vascular disorders) | 5 (5) — Symptomatic intracerebral hemorrhage
Perforation (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Acute Ischemic Stroke (N=60)
Asymptomatic hemorrhage (Vascular disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days